CLINICAL TRIAL: NCT01264523
Title: Short-term Effect of the Intake of Moderately High-protein, Low-glycemic Load Products on Anthropometrical, Glucose Metabolism and Lipid Metabolism Biomarkers, in Type-2 Diabetes Patients
Brief Title: Nutritional Intervention With Moderately High-protein, Low-glycemic Load Products in Type-2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Rovi Pharmaceuticals Laboratories (Industry); Equipe Enervit (Unknown)
Responsible Party: Principal Investigator, Alfredo Martinez, Main investigator, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UNAV-ROVI-001-2010
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Type-2 Diabetes; Overweight
Keywords: chrononutrition; moderately high protein; glycemic index; type-2 diabetes; overweight; obesity; weight management
MeSH Terms: conditions — Overweight; Obesity

INTERVENTIONS:
Other: Chronologically scheduled snacking with 40-30-30 products — Short-term analysis of the effects of the substitution of the habitual breakfast, mid-morning and afternoon snack of type-2 diabetes patients by 40-30-30 products. Longitudinal 2-period study
  Other Names: Enervit, Zone diet

SUMMARY:
The main objective of this study is to evaluate the effects on anthropometric, glucose metabolism and lipid profile biomarkers of exchanging with high-protein, low-glycemic index products (40-30-30) the habitual breakfast, mid-morning and afternoon snacks on type-2 diabetes patients following a chronologically scheduled pattern.

DETAILED DESCRIPTION:
Type 2 diabetes prevalence in adults has grown in the last years in many societies, accompanying the high incidence of obesity-related and other cardiovascular risk factors. Indeed, obesity is the most relevant overnutrition disease worldwide, being more dramatic than a self-esteem problem or an aesthetic issue, since it is associated to different metabolic disorders such as coronary diseases, hypertension, certain tumors, dislipidemia, biliary disorders, immunodeficiencies and insulin resistance. Different studies have shown the efficacy of low-fat diets on weight reduction, which has been associated to an improvement in overweight-related chronic pathological conditions. Additionally, a moderate increase of protein content (up to 30% of total caloric intake) in the diet and the inclusion of low-glycemic index products have been shown as a good tool for weight loss and maintenance. Recent studies have also shown the benefits of partial nutritional interventions, mainly on modifying breakfast intake, on anthropometrical and cardiovascular risk factors in overweight patients.

The study has been designed as a longitudinal nutritional intervention with two consecutive 4-week periods: from week 0 to 4, volunteers will follow their habitual diet. The second period (week 4 to 8), the volunteers' habitual breakfast, mid-morning and afternoon snacks will be substituted by 40-30-30 products, without changing any other parameter of their habitual diet or lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed of type-2 Diabetes
* Under dietary treatment or with Metformin
* Body Mass Index (BMI) Between 22 and 35 kg/m2

Exclusion Criteria:

* BMI under 22 or over 35 kg/m2
* To follow a pharmacological treatment with other drugs but metformin
* To be already insulin-dependent
* To have other concomitant pharmacological treatments for weight loss, hormonal substitutive therapy, altered thyroid function, etc. without an stable dosage (at least three months prior the beginning of the study).
* To suffer from complications due to type 2 diabetes (microangiopathy, polyneuropathy, cardiopathy, hepatic and renal impairments, etc)
* To have a recent (less than 3 months before the beginning of the study) uncontrolled diagnostic of hypercholesterolemia and/or hypertriglyceridemia.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Total Body weight | weeks 0, 4 and 8
  Total body weight will be measured at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
Fat Mass | weeks 0, 4 and 8
  Fat Mass will be measured at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
Fat-free mass | weeks 0, 4 and 8
  Fat-free mass will be measured at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).

SECONDARY OUTCOMES:
Hip circumference | weeks 0, 4 and 8
  Hip circumference will be measured at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
Waist circumference | weeks 0, 4 and 8
  waist circumference will be measured at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
Basal glucose concentration | weeks 0, 4 and 8
  Basal glucose concentration will be measured at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
Basal Insulin Concentration | weeks 0, 4 and 8
  Basal insulin concentration will be measured at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
HOMA-IR index | weeks 0, 4 and 8
  HOMA-IR index will be calculated based on basal glucose and insulin levels, at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
Glucose postprandial response | weeks 4 and 8
  Glucose concentrations will be analysed during the postprandial period after the habitual and the intervention breakfast intake at the end of both periods (weeks 4 and 8). Blood extractions will be performed at 0, 30, 60 and 120 minutes after the ingestion of the breakfasts
Insulin postprandial response | weeks 4 and 8
  Insulin concentrations will be analysed during the postprandial period after the habitual and the intervention breakfast intake at the end of both periods (weeks 4 and 8). Blood extractions will be performed at 0, 30, 60 and 120 minutes after the ingestion of the breakfasts
Basal Total Cholesterol | weeks 0, 4 and 8
  Total cholesterol concentration will be measured at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
HDL-Cholesterol | weeks 0, 4 and 8
  HDL-cholesterol concentration will be measured at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
Triglycerides Levels | weeks 0, 4 and 8
  Triglycerides concentration will be measured at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
LDL-cholesterol | weeks 0, 4 and 8
  LDL-cholesterol concentration will be calculated based on the FRiedewald Formula at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
C-Reactive Protein | weeks 0, 4 and 8
  C-Reactive Protein concentration will be measured at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
Homocystein | weeks 0, 4 and 8
  Homocystein concentration will be measured at the beginning of the study (week 0), at week 4 (before starting the intervention with 40-30-30 products) and week 8 (end of the study).
Dietary intake | during first period (week 0-4) and second period (week 4-8)
  Dietary intake will be evaluated through 72h food records, which will be filled by the volunteers during 3 days in the habitual intake period (week 0-4) and during the intervention period (week 4-8)
Satiety assessment | weeks 4 and 8
  During the postprandial period after the ingestion of the habitual breakfast (week 4) and the 40-30-30 breakfast (week 8), volunteers will fill a total of four Visual Analogue Scale (VAS) questionnaires, at times 0, 30, 60 and 120 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Martinez, PhD, Principal Investigator — University of Navarra; Santiago Navas-Carretero, PhD, Study Chair — University of Navarra; Itziar Abete, PhD, Study Chair — University of Navarra; M. Angeles Zulet, PhD, Study Chair — University of Navarra
Locations (1):
- Department of Nutrition, Food Science, Physiology and Toxicology. University of Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Result] Navas-Carretero S, Abete I, Zulet MA, Martinez JA. Chronologically scheduled snacking with high-protein products within the habitual diet in type-2 diabetes patients leads to a fat mass loss: a longitudinal study. Nutr J. 2011 Jul 14;10:74. doi: 10.1186/1475-2891-10-74. PMID 21756320
- See also: European Master´s Degree in Feeding, Nutrition and Metabolism — http://www.unav.es/master/nutricion-metabolismo/